CLINICAL TRIAL: NCT06073496
Title: The Effectiveness of Electroacupuncture and Standard Therapy Compared to Standard Therapy in Gynecological Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Zulaika Rosalin, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-06-0970
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Gynecologic Cancer; Cancer Related Pain; Cancer Pain
Keywords: Electroacupuncture; Cancer pain; Gynecological cancer pain; Acupuncture; VAS; EORTC QLQ C 30; Quality of Life; Analgetic Dose
MeSH Terms: conditions — Cancer Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: asessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Patient are cancer patient that experience cancer pain that only receive analgetic drug treatment according to WHO Stepledder of Pain
- Electroacupuncture and standard Therapy (Experimental): The Patient are cancer patient that experience cancer paint that receive analgetic drug treatement according WHO stepledder of pain and receive electroacupuncture
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Patient receive analgetic medicine will get experimental procedure with needle insertion that attach to eletrostimulator
  Arms: Electroacupuncture and standard Therapy

SUMMARY:
Gynecological cancer is cancer that starts in the female reproductive organs. Pain in gynecological cancer can be caused by an underlying malignancy or surgical procedure as well as chronic pain associated with malignancy and sequelae of the therapy given. Gynecological cancer patients often experience moderate to severe pain and use higher levels of opioids than patients diagnosed with other cancers. More than two thirds of patients with advanced cancer experience severe pain and up to half of these patients report that their pain is not well controlled. This study aims to analyze the effectiveness of electroacupuncture plus standard therapy on pain intensity (VAS score), changes in analgesic dose, and quality of life (QLQ C-30 EORTC score) in patients with gynecological cancer pain compared to standard therapy alone.

DETAILED DESCRIPTION:
This study was conducted using single blinded randomized control clinical trial, design in 58 patients diagnosed with gynecological cancer, aged 18 to 65 years, who experienced cancer pain, with VAS ≥ 4, pain caused by a tumor, before or while undergoing a therapeutic process (radiation therapy, chemotherapy, or post surgery), side effects or due to the toxicity of cancer treatment, willing to take part in this study and sign informed consent who were randomized into 2 groups, namely group I electroacupuncture with standard therapy and group 2 standard therapy, the acupuncture points used were LI4, PC6, ST36, SP6 and LR3, after the acupuncture needle was inserted, the needle was connected to the electrosimulator. The outputs assessed were pain intensity using the VAS, changes in analgesic dose, and quality of life with the EORTC QLQ C-30 questionnaire, which was assessed on the day before starting therapy, the first day, the second day, the third day, the fifth day and the seventh day.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 to 65 years old
* Gynecocal cancer with pain ≥ 4 acording Visual Analog scale and receive analgetic medicine
* The pain cause by

  1. direct from cancer
  2. Treatment proces surgery, radiotherapy, chemotherapy, paliatif treatment, supportive treatment
  3. Adverse reaction form treatment and intoxication

Exclusion Criteria:

* Emergency case patient with hemodynamic instable
* Patient with uncooperative behavior because ith serious psychological disorders, no currently undergoing psychiatric treatment, aggressive behavior, that not allowed for acupuncture.
* Patients with blood clotting disorders, with platelets <50.000 and in neutropenic condition with <1000 neutrophils.
* The patient has an allergy to stainless steel acupuncture needles. Wounds at the acupuncture point puncture sites, skin infections in the ears. On patients with eczema on the ears, external otitis or psoriasis.
* There is a tumor in the area that will be stabbed and stimulated in the stomach pregnant women, close to the heart, or in the area of the carotid sinus lymphedema, insertion into the prosthesis.
* Patients with heart rhythm disorders. The patient uses a pace maker.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with gynecology cancer
Enrollment: 58 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Pain severity with Visual Analog Scale | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  Rating scale for measuring pain, where the minimum value is 0 = no pain, and the maximum value is 100 = severe pain. A higher scale means worse outcomes.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life C30 | before treatment and 7 day after treatment
  A Quesionaire for measuring quality of Life
Analgetic Usage in dosage and frequency | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  by assessing drug dose reductions and frequency before and after

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia
Locations (3):
- Indonesia (3):
  - Fatmawati Hospital, Jakarta, DKI Jakarta
  - Persahabatan Hospital, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No